# Effect of Aldosterone on Myocardial Energy Starvation

NCT00574119

February 22, 2011

Effect of Aldosterone on Myocardial Energy Starvation

Marvin W. Kronenberg, M.D.

Version 6 Revised February 22, 2011

#### PROPOSED RESEARCH PLAN

This proposal is intended to obtain sufficient data to allow an application to the NHLBI to further our understanding of the pathophysiology of heart failure (HF) and to evaluate the "energy starvation hypothesis" of HF in patients. We can now use metabolic imaging with positron emission tomography (PET) and anatomic-functional imaging with cardiac magnetic resonance (CMR) to study energy starvation in HF.

# 1. SPECIFIC AIMS:

- a. To employ PET and CMR to evaluate several determinants of myocardial "energy starvation" in patients with HF due to nonischemic dilated cardiomyopathies (NIDCM):
  - 1) Left ventricular (LV) volume, ejection fraction (LVEF) and wall stress (CMR).
  - 2) LV hypertrophy (LVH) and fibrosis (CMR).
  - 3) LV subendocardial hypoxia, using blood oxygen level derived (BOLD) imaging and adenosine/regadenoson-induced hyperemia imaging (CMR).
  - 4) The rate of myocardial oxidative metabolism using [11C]acetate (PET).
- b. To study LV energy supply-demand relations and efficiency in patients with NIDCM using the [11C]acetate decay rate, kmono, an index of energy supply, compared to indices of demand (LV wall stress and the rate-pressure product) plus an index of efficiency, the work-metabolic index (LV minute work/kmono).
- c. To evaluate LV mass, volume and LVEF before and after aldosterone blockade, compared to changes in myocardial fibrosis, reactive hyperemia, BOLD estimates of hypoxia and myocardial oxidative metabolism.
- d. To evaluate the relations between clinical improvement, energy starvation and LV volume, for judging the hypothesis that drugs that reduce LV fibrosis and volumes are beneficial in HF.
- e. To evaluate the reproducibility of CMR measurements of myocardial perfusion.
- **2. BACKGROUND AND SIGNIFICANCE:** (References are sometimes listed, rather than discussed in detail, due to page limits.). **Energy starvation**. Heart failure (HF) may be caused by myocyte death, myocyte dysfunction and LV remodeling, leading to ischemia and neurohormonal abnormalities, with inadequate energy production, termed "energy starvation", with HF progression ( $^1$ ), key elements in the HF syndrome.( $^2$ , $^3$ ). **There are long term maladaptive anatomical responses related to energy starvation**, especially hypertrophy, reduced capillary density and abnormal mitochondrial architecture. **Energy-sparing compensation**. B-adrenergic downregulation is important, but is maladaptive by reducing LV performance, increasing  $\beta$ -myosin heavy chains and decreasing sarcoplasmic reticulum calcium pumping sites ( $^{1,3}$ ). **Remodeling** ( $^4$ , $^5$ , $^6$ , $^7$ , $^8$ , $^9$ , $^{10}$ , $^{11}$ , $^{12}$ ). Remodeling includes LV dilation, LVH and reduced function. There is reexpression of fetal gene programs ( $^{9,10}$ ). Myocyte loss (via necrosis and apoptosis) leads to subendocardial cell death with replacement fibrosis and a loss of vasodilator reserve ( $^{12}$ ) (all related to poorer prognosis).

Aldosterone and myocardial fibrosis. Aldosterone's (ALDO) role in LV pathology and HF became clearer following publications showing neurohormonal profiles in HF (13,14) and research showing the reninangiotensin-aldosterone system was related to LVH and fibrosis (15,16,17,18). Two HF trials showed reduced mortality in patients with HF randomized to treatment with the ALDO antagonist, spironolactone (19), or eplerenone (20) following myocardial infarction. A substudy of RALES showed decreased B-type natriuretic peptide (BNP) in patients randomized to spironolactone (21). Tsutamoto found in patients a decrease by spironolactone of the myocardial extraction of ALDO (22). In a randomized study of patients with NIDCM and H, 4 months' treatment of 20 patients with spironolactone was associated with significantly reduced LV mass and volume, increased LVEF, and neurohormonal improvements, with a decrease in BNP, plus a decrease in plasma procollagen type III aminoterminal peptide (PIIINP) (23), an index of myocardial fibrosis. Decreased LV mass on echocardiography was correlated with decreased PIIINP. Others confirmed a slight increase in LVEF with spironolactone in HF patients (24,25). In animals with myocardial infarctions, eplerenone increased the speed of isovolumic relaxation, increased endothelial nitric oxide synthase, and also reduced type I collagen gene expression and LVH (26). Similarly, eplerenone reduced LV hydroxyprolene, improved LV filling and

coronary blood flow dynamics in the spontaneously hypertensive rat (<sup>27</sup>). Noncardiac mechanisms involve blockade of brain mineralocorticoid receptors leading to reduced sympathetic outflow and improved cardiac function in the rat following MI (<sup>28</sup>). Thus, there is substantial clinical evidence of cardiac benefit from ALDO blockade, confirmed in rat models, but relatively little evidence in patients for an actual reduction in fibrosis, or other mechanisms of benefit. We speculate that ALDO blockade in patients with HF will reduce fibrosis and LV mass, which will likely reduce LV diastolic pressure and likely improve subendocardial perfusion, leading to less subendocardial ischemia in HF. This would improve the anatomic and physiologic substrate of "energy starvation".

Oxidative metabolism and cardiac efficiency in HF. Several studies have examined oxidative metabolism and LV efficiency in patients with HF, both using catheterization techniques (<sup>29</sup>) and noninvasive methods that employ PET and echocardiography (<sup>30</sup>, <sup>31</sup>, <sup>32</sup>). Oxidative metabolism can be estimated from the rate of clearance of [<sup>11</sup>C]acetate from myocardium (kmono), which correlates closely with myocardial oxygen consumption (MVO2) in animal models (<sup>33</sup>, <sup>34</sup>, <sup>35</sup>). Importantly, in NIDCM patients there is a similar, quantitative linear relation between [<sup>11</sup>C]acetate decay and LV oxygen consumption (<sup>30</sup>). Efficiency may be judged by the work-metabolic index (WMI) = LV minute work/kmono. WMI has improved following metoprolol (<sup>36</sup>), but this has not yet been related to the anatomical substrate of energy starvation or to changes in that substrate.

Cardiac magnetic resonance imaging (CMR). CMR has become a "gold standard" method for cardiac imaging. There is a quantitative relation of CMR to LV mass, volume and performance (37,38) and it is highly reproducible (39). CMR is likely to be superior to echocardiography in judging the work-metabolic index. Imaging LV vasodilator reserve and hypoxia with CMR. Panting et al recently used gadolinium with adenosine/ regadenoson to image marked, inadequate subendocardial perfusion (40). Deoxyhemoglobin is paramagnetic (41) and can be seen on BOLD images. Several studies have employed this property to study hypoxia and ischemia (41,42,43,44,45,46,47,48). There is a blunted dipyridamole-induced change in the BOLD transverse relaxation rate with LVH (p=0.0003), although in this study, none had HF (47). It is important to note the distinction between hypoxia and ischemia. BOLD shows deoxyhemoglobin, but by itself cannot differentiate hypoxia from ischemia induced by hypoxia. Inducible LV dysfunction associated with a large BOLD signal would be confirmatory evidence, but is not likely to be proven in this study, as

opposed to study of patients with coronary artery disease.

Critical evaluation of existing knowledge, gaps which this project is intended to fill, importance and relevance of the proposed research. We hope to demonstrate in patients several anatomic and physiologic abnormalities that produce myocardial "energy starvation" in HF, and that energy starvation is reduced by therapy with the ALDO antagonist, spironolactone. Gaps in our knowledge include: 1) Most basic information regarding ALDO has been obtained in animal models, whereas clinical reports have mostly shown cruder information such as reduced LVH and improved LVEF (cited above). 2) No clinical studies have addressed specifically the substrate of energy starvation in HF. 3) To our knowledge, there is no information about whether ALDO antagonism can reverse subendocardial hypoxia, and possibly ischemia, and only partial information in patients about fibrosis from serum markers, such as PIIINP 4) There is little mechanistic information to add physiologic support for the volume-remodeling hypothesis of how drugs improve outcomes in HF. 5). There are no reproducibility data regarding resting or adenosine-stimulated myocardial blood flow using CMR.

This study is likely to reduce these gaps in our knowledge of HF. By CMR and PET, we expect to show "energy starvation" in NIDCM by demonstrating LVH and fibrosis, inadequate vasodilator reserve, hypoxia and reduced metabolism vs. demand. Treatment with spironolactone will allow study of the effects of this proven therapy on the anatomy and physiology of energy starvation. This will demonstrate the physiologic basis of the volume-remodeling hypothesis about how drugs improve outcomes in patients with HF. BOLD and [11C]acetate imaging may identify patients with the worst physiologic consequences of HF. Drug therapy, and even selection for cardiac transplantation, might be improved by this work. By doing repeated studies in a subset of patients, we expect to document close reproducibility of CMR estimates of myocardial perfusion. This will allow us to judge with greater confidence the serial changes we expect following spironolactone treatment.

**3. PRELIMINARY STUDIES BY APPLICANT:** The PI has studied HF in several formats (<sup>49</sup>, <sup>50</sup>, <sup>51</sup>, <sup>52</sup>, <sup>53</sup>) and recently completed a study of LV oxidative metabolism using PET, RPP and echocardiography in patients with NIDCM (figs 1-4) (<sup>54</sup>). Data for calculating kmono in NIDCM are shown in fig. 1. Compared to normal subjects, the LV supply/demand relation (kmono/RPP) was depressed in patients with NIDCM (fig 2). Normal subjects had a linear, significant relation between kmono and RPP, but patients with NIDCM did not (fig 3). Three of 7 patients had results similar to 7 normal subjects, but 4 did not. The literature demonstrates normally linear relations between LV wall stress and MVO2 (<sup>55</sup>, <sup>56</sup>). But, in the present study, there was no significant relationship in NIDCM between kmono and LV wall stress, as another index of oxygen demand (fig.4).





Fig. 1. Fig. 2.





Fig. 3. Fig. 4.

Such lack of correlation supports the hypothesis of "energy starvation" in HF. The PI has studied LV remodeling as part of the Radionuclide Substudy of SOLVD which was among the first to establish that the angiotensin converting-enzyme inhibitor, enalapril, reduced LV volume, while placebo-treated patients had progressive LV volume dilation (remodeling) (51). A meta-analysis showed that drugs that are clinically beneficial for HF reduce or have a neutral effect on LV volume (57). The PI has continued studies of the LV volume-remodeling hypothesis (58), used the 6 minute walk test (59) and has significant nuclear cardiology experience (please see biosketch).

# 4. RESEARCH DESIGN AND METHODS:

**Patient inclusion criteria.** We plan to study 10 patients with NIDCM in each of two years (n based on budget). Most patients will have hypertensive or idiopathic dilated cardiomyopathy. The limited literature suggests that with 20 patients we will see a significant improvement in LV ejection fraction(<sup>23</sup>).

The inclusion criteria are:

- 1) 18-80 years old, of either sex and any race;
- 2) diagnosis of NIDCM based on clinical criteria;
- 3) New York Heart Association Functional Class (NYHA FC) II-IV;
- 4) an ECG showing no prior myocardial infarction;

- 5) LV ejection fraction of 35% or less;
- 6) able to lie supine for PET and MRI studies.
- 7) standard medical therapy for heart failure, including an angiotensin converting enzyme inhibitor or an angiotensin receptor blocking drug; beta-adrenergic blocking drugs, and possibly digitalis and potassium, if needed; a no added salt diet; fluid restriction if needed. Patients will be stable on the above anit-failure therapy for 3 months.
- 8) Serum potassium less than 5.0 and serum creatinine 2.5 or less.

**Exclusion criteria** will include 1) need for an internal cardioverter-defibrillator (ICD) based on ventricular tachyarrhythmias (we cannot perform CMR in patients with ICD's); 2) other severe, concomitant illness; 3) prior stroke or orthopedic problems that limit exercise capacity. 4) Abnormal renal function as defined above; **Cautious exclusion**: For patients with chronic moderate obstructive pulmonary disease (COPD) of severity that requires chronic, daily inhaler therapy the physician may consider Regadenoson for the diagnostic portions of the MRI. This will be based on the physicians medical opinion. If the patient has severe COPD he/she will be excluded from the study.

**Recruitment Plan.** Patients with newly identified HF due to NIDCM will be recruited from Vanderbilt University Medical Center, the Nashville VA Medical Center and Meharry Medical College. After stabilization with the above treatments, we will request their participation in this study. Informed consent will be obtained using forms approved by our IRB.

# **CMR** Timeline





The above figures demonstrate the **protocol for the CMR and PET studies**. **For CMR**, patients will be studied while fasting to reduce chances of nausea during adenosine/regadenoson infusion. The HR and BP by sphygmomanometer will be recorded every minute during the adenosine/regadenoson infusion, and at least 5

times during the PET study. These results will be averaged. **For PET**, after an attenuation CT scan, kmono will be assessed with serial imaging after bolus injection of [¹¹C]acetate. The CMR and PET studies will be performed on the same day to reduce variability in BP, HR and medications between studies. Following PET, the patients will perform a 6-minute walk test 3 times for reproducibility within 10% of each other, with results on a standard form.

**Spironolactone therapy.** The initial dose will be 12.5 mg daily, and will be increased to 50 mg daily based on serum potassium and side effects, which will be monitored on days 3,7, 30 and then monthly. The BP, HR, body weight, cardiac physical examination, electrolytes and NYHA FC will be recorded at each visit on a standard form. If there is symptomatic gynecomastia with spironolactone, eplerenone, 25 or 50 mg as tolerated, will be used instead. **(20). Follow-up tests.** After 6 months' treatment, all the above tests will be repeated.

The following chart shows the protocol in table format.

| | Procedures for Aldo | sterone Study | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Screen and Consent | | Study<br>1 | | | | Study 2 | Study 2a |
| WEEK | 1 | 1.5 | 2 | 4 | 5 | 12 | 24 | 25 |
| History and Physical Exam | X | X | | X | X | X | X | |
| Spironolactone Dose | 25 | 25, CHK BMP, stop | 25 | 50 | | | | |
| Review Meds | X | X | X | X | X | X | X | |
| Basic Metabolic Panel (blood test) | X | X | X | X | X | X | X | |
| Blood Sampling for Heart Failure | | | X | | | | X | |
| 6 Minute Walking Test | | | X | | | | X | |
| Heart Failure Questionnaire | | | X | | | | X | |
| PET | | | X | | | | X | |
| CMR | | | X | | | | X | X |
| | UDY 1 AND 2 = the tests shown pasic metabolic profile to check p | | ion | | | | | |
| Sp | ironolactone dose may be adjust | ed up or down as needed | | | | | | |
| | Eplerenone may substitute t | for spironolactone | | | | | | |
| Wee | ks 1 and 5 may be done by draw | ring blood at other location | | | | | | |
| | Week 12 visit may be done by | telephone follow up | | | | | | |
| PET | $\Gamma$ = positron emission tomograph | y test of heart metabolism | | | | | | |

**Data analysis.** All results will be stored securely. PET and CMR data will be analyzed without reference to clinical data, and clinical results will be analyzed separately from CMR and PET data until finalized.

CMR = magnetic resonance imaging test of heart function, blood flow and scar tissue

Specific Aims a and b: Determinants of myocardial energy starvation, LV energy supply-demand relations and efficiency. With CMR we will accurately determine LVEDV, ESV, SV, LVEF and LV mass and calculate LV systolic wall stress with standard equations (60). Myocardial fibrosis will be graded using a visual, segmental method as outlined by McCrohon (61) in two representative short axis midventricular sections, with

results averaged. Myocardial reactive hyperemia will be estimated using gadolinium during adenosine/regadenoson infusion, according to the method of Panting ( $^{40}$ ). We will calculate percent voxels with inadequate reactive hyperemia. We will evaluate hypoxia using the BOLD imaging method suggested by Wacker ( $^{48}$ ) and will estimate the extent of myocardial hypoxia, according to the equation: [BOLD + voxels/Total voxels] x 100% = % BOLD + voxels. Lacking a predominantly subendocardial signal, we will employ a parametric analysis ( $^{62}$ ). Based on the findinds of Panting (40), we will compare myocardial perfusion in patients with NIDCM and normals.

<u>Specific comparisons</u>. We will evaluate the argument that subendocardial hypoxia by BOLD imaging is related to subendocardial ischemia, and that the volume of subendocardial hypoxia is related to LVEF. For this we will study the **correlation between LVEF and the %BOLD + voxels**. We recognize that other influences on each myocyte will also affect global LVEF, but we suspect that BOLD + regions may relate to LVEF.

We will evaluate the argument that LVH is the substrate for subendocardial hypoxia by **comparison of the %BOLD + voxels to LVH in gm**. The relation of LVH, %BOLD + voxels and LVEF may be complex and may require a 3-dimensional display to express it satisfactorily.

We will use CMR perfusion imaging with and without adenosine to compare myocardial perfusion in patients with NIDCM to patients with structurally normal hearts. Based on CMR procedural logs, we estimate there are up to 20 patients with structurally normal hearts studied with CMR during adenosine infusion. We will review the electronic medical records of these possible normal patients to determine if they have structurally normal hearts. We will then view and quantitatively analyze, using the method of Panting (40), these normal patients' images. We will compare the myocardial perfusion indices and myocardial perfusion reserve indices of the normals to that of patients with NIDCM.

We will **compare LV mass to the percent fibrosis** and will **evaluate the relation between fibrosis and \*BOLD + voxels** using standard linear correlation. We will quantify the monoexponential [11C]acetate decay rate using methodology we employed previously, averaging the [11C]acetate data in 4 midventricular slices.

<u>We will compare oxidative metabolic supply as estimated by kmono to 2 indices of myocardial demand, the RPP and LV systolic wall stress</u>. We expect this will confirm our prior, more limited observations, shown in the Preliminary Studies and will support the hypothesis of energy starvation in HF. We will calculate the WMI and compare this to results in the literature using the equation: WMI = (SBP x SVI x HR)/kmono, where SBP = systolic blood pressure, SVI = stroke volume index, HR = heart rate.

Specific Aim c: To evaluate relations among LV mass, volume and LVEF before and after aldosterone blockade, compared to changes in myocardial fibrosis, reactive hyperemia, BOLD estimates of hypoxia and myocardial oxidative metabolism. The improvements in clinical status, LV mass and LVEF have been shown in two studies, and we expect the same results. The goal of this Specific Aim is to judge the parameters of energy starvation (LVH, fibrosis, reactive hyperemia, LV hypoxia and oxidative metabolism) before and during 4 months' spironolactone treatment. Thus, we will compare changes in LVH, % fibrosis, %BOLD+ voxels and the percent reactive hyperemia to LVEDV, LVESV, LVEF, SV, kmono/RPP and the WMI before and during spironolactone treatment.

Specific Aim d: To evaluate the relations between clinical improvement, the energy starvation theory and LV volume, for judging the hypothesis that drugs that reduce LV volumes are beneficial in HF. We expect a spectrum of responses to aldosterone-blocking therapy. It will be useful to compare the response clinically and by LV volume analysis to myocardial supply-demand relations, BOLD imaging and reactive hyperemia. We will compare changes in LVEDV, LVESV, SV and LVEF to NYHA FC, 6-minute walk test performance to kmono/RPP, WMI, %BOLD+ voxels and reactive hyperemia. We will use paired t-tests and linear correlation. We believe these results will add evidence to support the volume-remodeling hypothesis.

**Specific Aim e. To evaluate the reproducibility of CMR measurements of myocardial perfusion.** We expect close reproducibility of the CMR estimates of myocardial perfusion at rest and during adenosine infusion, but since we have been unable to document this in the literature, we propose to perform this study in a subset of 8 HF patients. This is based on the advice of our biostatistical consultants. We will then have greater confidence in judging the changes that we expect to detect following spironolactone therapy.

Statistical analysis. Based on the only available actually randomized data ( $^{23}$ ) 20 subjects will provide statistically significant information for our goals. Subsequent NHLBI applications will have more detailed goals. The study of patients before and during spironolactone treatment will allow us to use each patient as his/her own control. The data analysis will employ standard techniques, including paired t-tests and linear regression analysis as appropriate. Statistical significance will be judged as p < 0.05.

Potential difficulties and limitations. Patient recruitment. We are confident it will be possible to recruit sufficient patients with NIDCM at Vanderbilt and the adjacent Nashville VA Medical Center. [¹¹C]acetate decay in HF. There is a strong, quantitative relation between myocardial oxygen consumption and [¹¹C] acetate decay in HF (³⁰). Thus, this measurement reflects oxidative metabolism in HF. BOLD and reactive hyperemia in HF. There is support in the literature (see Background) for making these measurements with our equipment (1.5 T magnet). Selection of spironolactone. The literature supports using this drug in HF(¹⁰) unless there are significant side effects of gynecomastia, whereupon we will change to eplerenone (²⁰). Timing of repeat testing. Based on the initial studies of spironolactone in NIDCM (²³) we expect to see by 4 months an improvement in LVEF and a decrease in LVEDV. Responders and nonresponders to spironolactone. We expect a spectrum of response to spironolactone. This should be a strength of the analysis of our data concerning the anatomic and physiologic mechanisms of energy starvation. A sample size of 20 patients (²³) should be adequate to demonstrate striking responses in some patients and to produce sufficient encouraging data for an application for further support

**5. ETHICAL ASPECTS OF THE PROPOSED RESEARCH:** We believe there are no ethical problems in the proposed research. Given the **well-documented benefits of ALDO-blocking drugs**, it is no longer ethical to conduct a placebo-controlled study of ALDO-blocking effects. Thus, we will use a before and after (during) approach. The problem of **when to implant an ICD** might be considered an issue. However, it is reasonable to institute aldo-blocking therapy, in addition to the other anti-failure therapy in newly diagnosed HF patients because this may improve LVEF such that an ICD may not be needed. **Present guidelines (63) are moot on the duration of treatment before placing an ICD**. However, If we discover significant ventricular arrhythmias during this research that require an ICD, we will end the patient's participation in the study and promptly notify the patient's physician of these developments. **Human subjects:** Consent will be obtained using forms approved by the Vanderbilt IRB. Women and minorities will be included. The targeted enrollment will be 20 subjects of both sexes for reasons noted above. Inclusion and exclusion criteria were listed above.

# LITERATURE CITED:

\_

<sup>&</sup>lt;sup>1</sup> Colucci WS and Braunwald EB. Pathophysiology of heart failure. In:Braunwald's Heart Disease. A Textbook of Cardiovascular Medicine. Zipes DP, Libby P, Bonow RO, Braunwald E, eds. 7th ed. Elsevier Saunders, Philadelphia, 2005. pp 512-524.

<sup>&</sup>lt;sup>2</sup> Ingwall JS, Weiss RG. Is the failing heart energy starved? On using chemical energy to support cardiac function. Circ Res. 2004;95:135-45.

<sup>&</sup>lt;sup>3</sup> Katz AM. Cardiomyopathy of overload. A major determinant of prognosis in congestive heart failure. N Engl J Med. 1990;322:100-10.

<sup>&</sup>lt;sup>4</sup> Sabbah HN, Sharov V, Riddle JM, Kono T, Lesch M, Goldstein S. Mitochondrial abnormalities in myocardium of dogs with chronic heart failure. J Mol Cell Cardiol. 1992;24:1333-47.

<sup>&</sup>lt;sup>55</sup> Unverferth DV, Leier CV, Magorien RD, Croskery R, Svirbely JR, Kolibash AJ, et. al. Improvement of human myocardial mitochondria after dobutamine: a quantitative ultrastructural study. J Pharmacol Exp Ther. 1980;215:527-32.

- <sup>9</sup> Dorn GW 2nd, Mann DL. Signaling pathways involved in left ventricular remodeling: summation. J Card Fail. 2002;8:S387-8.
- <sup>10</sup> Cohn JN, Ferrari R, Sharpe N. Cardiac remodeling--concepts and clinical implications: a consensus paper from an international forum on cardiac remodeling. On Behalf of an International Forum on Cardiac Remodeling. J Am Coll Cardiol. 2000;35:569-82.
- <sup>11</sup> Vatner SF. Reduced subendocardial myocardial perfusion as one mechanism for congestive heart failure. Am J Cardiol. 1988;62:94E-98E.
- <sup>12</sup> Neglia D, Michelassi C, Trivieri MG, Sambuceti G, Giorgetti A, Pratali L, et. al. Prognostic role of myocardial blood flow impairment in idiopathic left ventricular dysfunction. Circulation. 2002;105:186-93.
- <sup>13</sup> Benedict CR, Francis GS, Shelton B, Johnstone DE, Kubo SH, Kirlin P, Nicklas J, Liang CS, Konstam MA, Greenberg B, et al. Effect of long-term enalapril therapy on neurohormones in patients with left ventricular dysfunction. SOLVD Investigators. Am J Cardiol. 1995;75:1151-7.
- <sup>14</sup> Francis GS, Benedict C, Johnstone DE, Kirlin PC, Nicklas J, Liang CS, Kubo SH, Rudin-Toretsky E, Yusuf S. Comparison of neuroendocrine activation in patients with left ventricular dysfunction with and without congestive heart failure. A substudy of the Studies of Left Ventricular Dysfunction (SOLVD). Circulation. 1990;82:1724-9.
- <sup>15</sup> Brilla CG, Rupp H, Maisch B. Effects of ACE inhibition versus non-ACE inhibitor antihypertensive treatment on myocardial fibrosis in patients with arterial hypertension. Retrospective analysis of 120 patients with left ventricular endomyocardial biopsies. Herz. 2003;28:744-53.
- <sup>16</sup>Wilke A, Funck R, Rupp H, Brilla CG. Effect of the renin-angiotensin-aldosterone system on the cardiac interstitium in heart failure. Basic Res Cardiol. 1996;91 Suppl 2:79-84.
- <sup>17</sup> Brown NJ. Aldosterone and end-organ damage. Curr Opin Nephrol Hypertens. 2005;14:235-41. Weber KT. Aldosterone in congestive heart failure. N Engl J Med. 2001;345:1689-97.
- <sup>18</sup> Weber KT. Aldosterone in congestive heart failure. N Engl J Med. 2001;345:1689-97.
- <sup>19</sup> Pitt B, Zannad F, Remme WJ, Cody R, Castaigne A, Perez A, Palensky J, Wittes J. The effect of spironolactone on morbidity and mortality in patients with severe heart failure. Randomized Aldactone Evaluation Study Investigators. N Engl J Med. 1999;341:709-17.
- <sup>20</sup> Pitt B, Remme W, Zannad F, Neaton J, Martinez F, Roniker B, Bittman R, Hurley S, Kleiman J, Gatlin M; Eplerenone Post-Acute Myocardial Infarction Heart Failure Efficacy and Survival Study

<sup>&</sup>lt;sup>6</sup> Maytin M, Colucci WS. Molecular and cellular mechanisms of myocardial remodeling. J Nucl Cardiol. 2002;9:319-27.

<sup>&</sup>lt;sup>7</sup> Sawyer DB, Siwik DA, Xiao L, Pimentel DR, Singh K, Colucci WS. Role of oxidative stress in myocardial hypertrophy and failure. J Mol Cell Cardiol. 2002;34:379-88.

<sup>&</sup>lt;sup>8</sup> Hunter JJ, Chien KR. Signaling pathways for cardiac hypertrophy and failure. N Engl J Med. 1999;341:1276-83.

Investigators. Eplerenone, a selective aldosterone blocker, in patients with left ventricular dysfunction after myocardial infarction. N Engl J Med. 2003;348:1309-21.

- <sup>21</sup> Rousseau MF, Gurne O, Duprez D, Van Mieghem W, Robert A, Ahn S, Galanti L, Ketelslegers JM; Belgian RALES Investigators. Beneficial neurohormonal profile of spironolactone in severe congestive heart failure: results from the RALES neurohormonal substudy. J Am Coll Cardiol. 2002;40:1596-601.
- <sup>22</sup> Tsutamoto T, Wada A, Maeda K, Mabuchi N, Hayashi M, Tsutsui T, Ohnishi M, Sawaki M, Fujii M, Matsumoto T, Horie H, Sugimoto Y, Kinoshita M. Spironolactone inhibits the transcardiac extraction of aldosterone in patients with congestive heart failure. J Am Coll Cardiol. 2000;36:838-44
- <sup>23</sup> Tsutamoto T, Wada A, Maeda K, Mabuchi N, Hayashi M, Tsutsui T, Ohnishi M, Sawaki M, Fujii M, Matsumoto T, Matsui T, Kinoshita M. Effect of spironolactone on plasma brain natriuretic peptide and left ventricular remodeling in patients with congestive heart failure. J Am Coll Cardiol. 2001;37:1228-33.
- <sup>24</sup> Cicoira M, Zanolla L, Rossi A, Golia G, Franceschini L, Brighetti G, Marino P, Zardini P. Long-term, dose-dependent effects of spironolactone on left ventricular function and exercise tolerance in patients with chronic heart failure. J Am Coll Cardiol. 2002;40:304-10.
- <sup>25</sup> Feola M, Menardi E, Ribichini F, Vado A, Deorsola A, Ferrero V, Visconti G, Milanese U, Uslenghi E. Effects of the addition of a low dose of spironolactone on brain natriuretic peptide plasma level and cardiopulmonary function in patients with moderate congestive heart failure. Med Sci Monit. 2003;9:CR341-5.
- <sup>26</sup> Fraccarollo D, Galuppo P, Hildemann S, Christ M, Ertl G, Bauersachs J. Additive improvement of left ventricular remodeling and neurohormonal activation by aldosterone receptor blockade with eplerenone and ACE inhibition in rats with myocardial infarction. J Am Coll Cardiol. 2003;42:1666-73.
- <sup>27</sup> Susic D, Varagic J, Ahn J, Matavelli L, Frohlich ED. Long-term mineralocorticoid receptor blockade reduces fibrosis and improves cardiac performance and coronary hemodynamics in elderly SHR. Am J Physiol Heart Circ Physiol. 2007;292:H175-9.
- <sup>28</sup> Huang BS, Leenen FH. Blockade of brain mineralocorticoid receptors or Na+ channels prevents sympathetic hyperactivity and improves cardiac function in rats post-MI. Am J Physiol Heart Circ Physiol. 2005;288:H2491-7.
- <sup>29</sup> Eichhorn EJ, Heesch CM, Barnett JH, Alvarez LG, Fass SM, Grayburn PA, Hatfield BA, Marcoux LG, Malloy CR. Effect of metoprolol on myocardial function and energetics in patients with nonischemic dilated cardiomyopathy: a randomized, double-blind, placebo-controlled study. J Am Coll Cardiol. 1994;24:1310-20.
- <sup>30</sup> Beanlands RS, Bach DS, Raylman R, Armstrong WF, Wilson V, Montieth M, et. al. Acute effects of dobutamine on myocardial oxygen consumption and cardiac efficiency measured using carbon-11 acetate kinetics in patients with dilated cardiomyopathy. J Am Coll Cardiol. 1993;22:1389-98.
- <sup>31</sup> Beanlands RS, Armstrong WF, Hicks RJ, Nicklas J, Moore C, Hutchins GD, et. al. The effects of afterload reduction on myocardial carbon 11-labeled acetate kinetics and noninvasively estimated mechanical efficiency in patients with dilated cardiomyopathy. J Nucl Cardiol. 1994;1:3-16.

- <sup>35</sup> Armbrecht JJ, Buxton DB, Schelbert HR. Validation of [1-11C]acetate as a tracer for noninvasive assessment of oxidative metabolism with positron emission tomography in normal, ischemic, postischemic, and hyperemic canine myocardium. Circulation. 1990;81:1594-605.
- <sup>36</sup> Beanlands RS, Nahmias C, Gordon E, Coates G, deKemp R, Firnau G, et. al. The effects of beta(1)-blockade on oxidative metabolism and the metabolic cost of ventricular work in patients with left ventricular dysfunction: A double-blind, placebo-controlled, positron-emission tomography study. Circulation.2000;102:2070-5.
- <sup>37</sup> Myerson SG, Bellenger NG, Pennell DJ. Assessment of left ventricular mass by cardiovascular magnetic resonance. Hypertension. 2002;39:750-5.
- <sup>38</sup> Longmore DB, Klipstein RH, Underwood SR, Firmin DN, Hounsfield GN, Watanabe M, Bland C, Fox K, Poole-Wilson PA, Rees RS, et al. Dimensional accuracy of magnetic resonance in studies of the heart. Lancet. 1985;1:1360-2.
- <sup>39</sup> Grothues F, Smith GC, Moon JC, Bellenger NG, Collins P, Klein HU, Pennell DJ. Comparison of interstudy reproducibility of cardiovascular magnetic resonance with two-dimensional echocardiography in normal subjects and in patients with heart failure or left ventricular hypertrophy. Am J Cardiol.2002;90:29-34.
- <sup>40</sup> Panting JR, Gatehouse PD, Yang GZ, Grothues F, Firmin DN, Collins P, Pennell DJ. Abnormal subendocardial perfusion in cardiac syndrome X detected by cardiovascular magnetic resonance imaging. N Engl J Med. 2002;346:1948-53.
- <sup>41</sup> Pauling L, Coryell C. The magnetic properties and structure of hemoglobin. Proc Natl Acad Sci USA 1936;22:210-216.
- <sup>42</sup> Ogawa S, Lee TM, Nayak AS, Glynn P. Oxygenation-sensitive contrast in magnetic resonance image of rodent brain at high magnetic fields. Magn Reson Med 1990;14:68-78.
- <sup>43</sup> Ogawa S, Lee TM. Magnetic resonance imaging of blood vessels at high fields: in vivo and in vitro measurements and image simulation. Magn Reson Med 1990;16(1):9-18.
- <sup>44</sup> Wendland MF, Saeed M, Lauerma K, de Crespigny A, Moseley ME, Higgins CB. Endogenous susceptibility contrast in myocardium during apnea measured using gradient recalled echo planar imaging. Magn Reson Med. 1993;29:273-276.
- <sup>45</sup> Atalay MK, Reeder SB, Zerhouni EA, Forder JR. Blood oxygenation dependence of T1 and T2 in the iolated, perfused rabbit heart at 4.7T. Magn Reson Med. 1995;34:623-627.

<sup>&</sup>lt;sup>32</sup> Bengel FM, Permanetter B, Ungerer M, Nekolla S, Schwaiger M. Non-invasive estimation of myocardial efficiency using positron emission tomography and carbon-11 acetate--comparison between the normal and failing human heart. Eur J Nucl Med. 2000;27:319-26.

<sup>&</sup>lt;sup>33</sup> Brown M, Marshall DR, Sobel BE, Bergmann SR. Delineation of myocardial oxygen utilization with carbon-11-labeled acetate. Circulation. 1987:76:687-96.

<sup>&</sup>lt;sup>34</sup> Brown MA, Myears DW, Bergmann SR. Validity of estimates of myocardial oxidative metabolism with carbon-11 acetate and positron emission tomography despite altered patterns of substrate utilization. J Nucl Med. 1989;30:187-93.

- <sup>46</sup> Li D, Dhawale P, Rubin PJ, Haacke EM, Gropler RJ. Myocardial signal response to dipyridamole and dobutamine: demonstration of the BOLD effect using a double-echo gradient-echo sequence. Magn Reson Med. 1996;36:16-20.
- <sup>47</sup> Beache GM, Herzka DA, Boxermann JL, Post WS, Gupta SN, Faranesh AZ, Solaiyappan M, Bottomley PA, Weiss JL, Shapiro EP, Hill MN. Attenuated myocardial vasodilator response in patients with hypertensive hypertrophy revealed by oxygenation-dependent magnetic resonance imaging. Circulation. 2001;104:1214-1217.
- <sup>48</sup> Wacker CM, Hartlep AW, Pfleger S, Schad LR, Ertl G, Bauer WR. Susceptibility-sensitive magnetic resonance imaging detects human myocardium supplied by a stenotic coronary artery without a contrast agent. J Am Coll Cardiol 2003;41:834-840.
- <sup>49</sup> Kronenberg MW, Konstam MA, Edens TR, Howe DM, Dolan N, Udelson JE, Benedict C, Stewart D, Yusuf S for the SOLVD Investigators: Factors influencing exercise performance in patients with left ventricular dysfunction. *J Card Fail* 1998; 4: 159-167.
- <sup>50</sup> Konstam MA, Kronenberg MW, Udelson JE, Kinan D, Metherall J, Dolan N, Edens T, Howe D, Kilcoyne L, Benedict C, Youngblood M, Barrett J, Yusuf S: Effectiveness of preload reserve as a determinant of clinical status in patients with left ventricular systolic dysfunction. *Am J Cardiol* 1992; 69:1591-1595.
- <sup>51</sup> Konstam MA, Rousseau MF, Kronenberg MW, Udelson JE, Melin J, Stewart D, Nolan N, Edens TR, Ahn S, Kinan D, Howe DM, Kilcoyne L, Metherall J, Yusuf S, Pouleur H for the SOLVD Investigators: Effects of the angiotensin converting enzyme inhibitor, enalapril, on the long-term progression of left ventricular dysfunction in patients with heart failure. *Circulation* 1992; 86:431-438.
- <sup>52</sup> Konstam MA, Kronenberg MW, Rousseau MF, Udelson JE, Melin J, Stewart D, Dolan N, Edens TR, Ahn S, Kinan D, Howe DM, Kilcoyne L, Metherall J, Benedict C, Yusuf S, Pouleur H for the SOLVD Investigators: Effects of the angiotensin converting enzyme inhibitor, enalapril, on the long-term progression of left ventricular dilatation in patients with asymptomatic systolic dysfunction. *Circulation* 1993; 88:2277-2283.
- <sup>53</sup> Patten RD, Kronenberg MW, Benedict CR, Udelson JE, Kinan D, Stewart D, Yusuf S, Smith JJ, Kilcoyne L, Dolan N, Edens TR, Metherall J, Konstam MA: Acute and long term effects of the angiotensin-converting enzyme inhibitor, enalapril, on adrenergic activity and sensitivity during exercise in patients with left ventricular systolic dysfunction. *Am Heart J* 1997; 134: 37-43.
- <sup>54</sup> Kronenberg MW, Cohen GI, Leonen MF, Mladsi TA, Di Carli MF. Myocardial oxidative metabolic supply-demand relationships in patients with nonischemic dilated cardiomyopathy. J Nucl Cardiol. 2006;13:544-53.
- <sup>55</sup> Kissling G. Mechanical determinants of myocardial oxygen consumption with special reference to external work and efficiency. Cardiovasc Res. 1992;9:886-92.
- <sup>56</sup> Graham TP Jr, Covell JW, Sonnenblick EH, Ross J Jr, Braunwald E. Control of myocardial oxygen consumption: relative influence of contractile state and tension development. J Clin Invest. 1968;47:375-85.
- <sup>57</sup> Konstam MA, Udelson JE, Anand IS, Cohn JN. Ventricular remodeling in heart failure: a credible surrogate endpoint. J Card Fail. 2003;9:350-3.
- <sup>58</sup> Udelson JE, McGrew FA, Flores E, Ibrahim H, Katz S, Koshkarian G, O'Brien T, Kronenberg MW, Zimmer C, Orlandi C, Konstam MA. Multicenter randomized, double-blind, placebo-controlled study

on the effect of oral tolvaptan on left ventricular dilatation and function in patients with heart failure and systolic dysfunction. J Am Coll Cardiol 2007; in press.

- <sup>59</sup> Bittner V, Weiner DH, Yusuf S, Rogers WJ, McIntyre KM, Bangdiwala SI, Kronenberg MW, Kostis JB, Kohn RM, Guillotte M, et al. Prediction of mortality and morbidity with a 6-minute walk test in patients with left ventricular dysfunction. SOLVD Investigators. JAMA.1993;270:1702-7.
- <sup>60</sup> Reichek N, Wilson J, St John Sutton M, Plappert TA, Goldberg S, Hirshfeld JW. Noninvasive determination of left ventricular end-systolic stress: validation of the method and initial application. Circulation. 1982;65:99-108.
- <sup>61</sup> McCrohon JA, Moon JC, Prasad SK, McKenna WJ, Lorenz CH, Coats AJ, Pennell DJ.Differentiation of heart failure related to dilated cardiomyopathy and coronary artery disease using gadolinium-enhanced cardiovascular magnetic resonance. Circulation. 2003;108:54-9.
- <sup>62</sup> Beache GM, Herzka DA, Boxerman JL, Post WS, Gupta SN, Faranesh AZ, Solaiyappan M, Bottomley PA, Weiss JL, Shapiro EP, Hill MN.Attenuated myocardial vasodilator response in patients with hypertensive hypertrophy revealed by oxygenation-dependent magnetic resonance imaging. Circulation. 2001;104:1214-7.
- <sup>63</sup> Hunt SA; American College of Cardiology; American Heart Association Task Force on Practice Guidelines (Writing Committee to Update the 2001 Guidelines for the Evaluation and Management of Heart Failure). ACC/AHA 2005 guideline update for the diagnosis and management of chronic heart failure in the adult: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Update the 2001 Guidelines for the Evaluation and Management of Heart Failure). J Am Coll Cardiol. 2005;46:e1-82.